CLINICAL TRIAL: NCT07375745
Title: Combined Gait Training and Transcutaneous Spinal Cord Stimulation to Enhance Lower Limbs Motor Recovery After Subacute SCI
Brief Title: Spinal Stimulation With Gait Training to Improve Lower Limbs Motor Recovery in Spinal Cord Injury
Acronym: CIMELocomotion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRIR 2025-2082
Record Dates: First submitted 2025-12-23; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury Subacute; Locomotion; Gait Disorder, Sensorimotor; Gait Disorders
Keywords: Spinal Cord Injury; Neuromodulation; Locomotion; tSCS; Non-invasive; Transcutaneous; Gait; Transcranial Magnetic Stimulation; Subacute; Artificial Intelligence; AI; Lower Limb; Gait training; Walking; Transcutaneous spinal stimulation; Tonic stimulation; Combined gait training and neuromodulation
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Pragmatic double-blind randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gait training alone (n=20) (Sham Comparator): Participants with spinal cord injury (SCI) classified as AIS A-D will receive sham transcutaneous spinal cord stimulation (tSCS) combined with robotic-assisted, treadmill, or overground gait training. The sham stimulation will reproduce the sensory sensation of active tSCS without eliciting effective spinal activation, ensuring participant blinding.
  The type of gait training will be determined based on the severity of the injury and the participant's ability to generate voluntary or assisted locomotor movements. Each participant will complete 20 training sessions, delivered four times per week over approximately five weeks.
  The gait training sessions will be individualized and task-specific, emphasizing repetitive stepping practice to promote locomotor learning and engage spinal and supraspinal networks involved in walking.
  Interventions: Other: Protocol 1: Gait training combined with a sham stimulation
- Gait training + tSCS (n=20) (Experimental): Participants with spinal cord injury (SCI) classified as AIS A-D will receive active transcutaneous spinal cord stimulation (tSCS) combined with robotic-assisted, treadmill, or overground gait training. The stimulation intensity will be individually adjusted to facilitate voluntary movement generation and enhance activation of spinal circuits involved in locomotion.
  The type of gait training will be determined based on the severity of the injury and the participant's ability to generate locomotor movements. Each participant will complete 20 training sessions, delivered four times per week over approximately five weeks.
  The gait training sessions will be individualized and task-specific, emphasizing repetitive stepping practice to promote locomotor learning and engage spinal and supraspinal networks responsible for walking.
  Interventions: Other: Protocol 2: Gait training combined with an effective tSCS

INTERVENTIONS:
Other: Protocol 1: Gait training combined with a sham stimulation — The training will be conducted using either the G-EO System (ReHa Technology) or a treadmill/overground with participants secured by a bodyweight support system (Biodex) to reduce bodyweight and prevent falls. Participants will complete 20 training sessions over a periode of 5 to 6 weeks. Each session will last up to 40 minutes, with rest periods if needed in case of performance decline.
  Each session will begin with a warm-up phase (5 minutes) to evaluate the condition of the participant and to ensure safety. On the G-EO System, this consists of using Passive Mode, which fully compensates for the participant's motor deficits. On the treadmill, the warm-up involves full hand assistance to guide gait.
  In sham-group, participants will combined gait training with a sham stimulation sets at sensory threshold, providing the perception of stimulation without activating locomotor spinal circuits.
  Arms: Gait training alone (n=20)
Other: Protocol 2: Gait training combined with an effective tSCS — The training will be conducted using either the G-EO System (ReHa Technology) or a treadmill/overground with participants secured by a bodyweight support system (Biodex) to reduce bodyweight and prevent falls. Participants will complete 20 training sessions over a periode of 5 to 6 weeks. Each session will last up to 40 minutes, with rest periods if needed in case of performance decline.
  Each session will begin with a warm-up phase (5 minutes) to evaluate the condition of the participant and to ensure safety. On the G-EO System, this consists of using Passive Mode, which fully compensates for the participant's motor deficits. On the treadmill, the warm-up involves full hand assistance to guide gait.
  In experimental group, participants will combined gait training with tSCS at T11-L2, sets to individualized parameters determined to facilitate lower limbs movement generation.
  Arms: Gait training + tSCS (n=20)

SUMMARY:
Spinal cord injury (SCI) often results in partial or complete loss of movement. In the subacute phase (< 6 months), the central nervous system shows increased potential for neuroplasticity, making it more responsive to rehabilitation and external stimulation. Standard care in rehabilitation centers relies on activity-based therapy (ABT), which uses intensive, task-specific training to promote recovery. Although ABT can improve mobility, its effects are often limited due to the nature of SCI and the indirect activation of neural circuits.

Recent findings suggest that adding transcutaneous spinal cord stimulation (tSCS) to ABT in chronic SCI (> 12 months) can enhance lower-limb motor recovery. This study will evaluate whether combining tSCS with gait training is safe and feasible in individuals with subacute SCI and whether it improves lower-limb motor outcomes compared with gait training alone.

The investigators hypothesize that pairing gait training with tSCS early after injury will be safe and feasible and that tSCS delivered during gait training will augment leg muscle activation and lead to greater functional improvements. The study will also assess the feasibility, safety and tolerability of implementing this combined intervention in a intensive functional rehabilitation setting.

DETAILED DESCRIPTION:
This study is lead by Dorothy Barthélemy (Ph.D, pht, Principal Investigator) and Nicolas Hoang Quang (M.Sc, Ph.D student) and collaborators, Marina Martinez (Ph.D), Marco Bonizzato (Ph.D) and Diana Zidarov (Ph.D).

Spinal cord injury (SCI) often results in partial or complete loss of motor function, greatly impacting independence and quality of life. During the subacute phase of recovery, defined as the first 6 months after injury, the central nervous system enters a period of heightened neuroplasticity in which it becomes especially responsive to rehabilitation and external stimulation. This critical window offers an opportunity to maximize motor recovery through targeted interventions.

In rehabilitation centers, the current standard of care focuses on activity-based therapy (ABT). ABT consists of intensive, repetitive and task-specific exercises designed to activate neural circuits below the level of injury, strengthen spared pathways and promote the formation of new neural connections. Although ABT has demonstrated benefits, it is frequently insufficient to restore functional walking, even when delivered intensively. As part of the CIME (Clinic for Intensive and Neuromodulation for Individuals with Spinal Cord Injury) Program, this study aims not to remain passive observers of the participant's nervous system as it attempts to generate the sensory inputs required for motor recovery. Instead, the investigators aim to actively enhance these inputs through targeted neuromodulation.

Recent evidence in chronic SCI suggests that combining ABT with transcutaneous spinal cord stimulation (tSCS) may augment the activity of spinal circuits involved in movement. tSCS is a non-invasive form of electrical stimulation applied to the skin over the spine, capable of activating dorsal root afferents and increasing the excitability of spinal networks. In this study, tSCS is used to provide direct, patterned sensory input to the CNS to potentially improve motor output during gait training.

This pragmatic randomized clinical trial will evaluate the safety and feasibility of combining task-specific gait training-delivered using robotic-assisted gait devices, treadmill-based therapy, or overground walking, with tSCS delivered Neurotrac Myoplus (FDA-approved stimulator) beginning as early as 4 to 6 weeks post-injury, within an intensive functional rehabilitation program. The study will also examine whether the addition of tSCS enhances lower-limb motor recovery in individuals with subacute SCI compared with gait training alone.

The investigators hypothesize that delivering tSCS during gait training early after injury will be safe and feasible, and that the combined intervention will increase leg muscle activation and lead to greater functional improvements than gait training alone. Feasibility, safety and tolerability of the combined approach will be systematically assessed to inform future clinical applications and larger-scale trials.

ELIGIBILITY:
Inclusion Criteria:

* paraplegic or quadriplegic participants with a subacute spinal cord injury (sSCI), defined as the stage of spinal cord damage occuring between 1 week and 6 months post-injury
* above 16 years old
* have a lesion between C1 - L2
* be considered as AIS A to D
* be able to stay at least 10 minutes standing with or without assistance
* can provide informed consent (no cognitive deficits by MoCA)
* be able to follow instructions in French or English

Exclusion Criteria:

* pacemaker
* active cancer on stimulation site or metastatic cancer
* unhealed wound, scar or pain which makes positioning of the electrodes impossible
* participants with specific contraindications to TMS (epilepsy, non-union cranial fracture and increased intracranial pressure) will be able to participate in the study, but will not receive TMS
* chronic and severe neuropathic pain
* pharmacology or implants that may impede with rehabilitation or spinal stimulation
* pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Motor Score | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Lower Extremity Motor Score (LEMS), derived from the ASIA Impairment Scale, is scored from 0 to 50, with higher scores indicating better motor function.

SECONDARY OUTCOMES:
Transspinal evoked potentials | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  The transspinal evoked potentials (TEPs) are muscle responses (Soleus, Tibialis Anterior, Vastus Lateralis and Biceps Femoris) recorded by electromyography (EMG) after tSCS.
  For each muscle, the resting motor threshold (RMT), the lowest intensity to elicit a motor response, will be measured. Additionally, normalized TEPmax (TEPmax/Mmax ratio) will be calculated to quantify the proportion of the maximal muscle response elicited by tSCS relative to the maximal direct motor response (Mmax). This ratio provides an index of spinal excitability and the effectiveness of stimulation in activating motor circuits.
Cortical excitability | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Transcranial magnetic stimulation (TMS) over the motor cortex will be used to assess corticospinal tract excitability. The latency and amplitude of motor evoked potentials (MEPs), as well as the active and resting motor threshold of the Tibialis Anterior muscle, will be measured.
Muscle strength | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Muscle strength will be evaluated using a handheld dynamometer (MicroFET), with measurements expressed in kilograms (kg). Higher values indicate greater muscle strength. Nine movements will be tested bilaterally : hip abduction, hip extension, hip flexion, knee extension, knee flexion, ankle dorsiflexion, ankle eversion, ankle inversion and ankle plantarflexion.
Spasticity | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Spasticity in the lower limbs will be assessed after the intervention using the Modified Ashworth Scale by a trained physical therapist. The examiner will passively move the limb through its full range of motion at a constant speed and rate the resistance encountered. The test is scored on a 6-point ordinal scale ranging from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension), with higher scores indicating greater levels of spasticity.
Sensory function | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Sensory function will be assessed using the sensory component of the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI). Light touch and pinprick sensations will be tested bilaterally across key dermatomes and scored on an ordinal scale. The total sensory score ranges from 0 to 56 (each for light touch and pinprick), with higher scores indicating better preserved sensory function.
Sensory function (2) | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Light touch and protective sensation will be assessed using Semmes-Weinstein monofilaments. Monofilaments of varying thickness will be applied perpendicularly to specific sites on the plantar surface of the foot or other areas of interest, until the filament bends. Participants will indicate whether they can perceive the touch. Each site will be tested multiple times to ensure reliability. The presence of sensation at thinner filaments indicates better sensory function, whereas inability to detect thicker filaments suggests sensory loss.
Balance and trunk control | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Balance will be assessed using the Modified Functional Reach Test (MFRT). Participants will be asked to reach forward as far as possible without taking a step or losing their balance, while sitting. The distance (in centimeters) reached is measured from the starting position of the fingertips to the maximal forward reach. Each trial will be performed three times and the average distance will be recorded. Higher reach distances indicate better dynamic balance and postural stability.

OTHER OUTCOMES:
Somatosensory changes following gait training combined with tSCS using EEG | 3 time frames : At day 0 (= baseline, prior to the first training session), up to one week after day 20 (= the last training session) and one month after day 20
  Tibial nerve stimulation will be applied and responses will be recorded by electroencephalogram (EEG) prior to and following the intervention. Evaluation of the latency and amplitude of somatosensory evoked potential (SSEP) will be realized.
Evaluation of safety and feasibility | Throughout the entier duration of the participation : From day 0 to one month after day 20.
  The investigators aim to evaluate if combining transcutaneous spinal cord stimulation with task-specific gait training is feasible early after the lesion is safe and feasible.
  For safety, the investigators are going to monitored adverse events and all participants will fill a qualitative questionnaire. This questionnaire will notably evaluate how the participant felt safe during the whole study (assessments and training sessions). Feasibility is assessed through recruitment and retention rates, % completion of expected number of sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de réadaptation Gingras-Lindsay-de-Montréal (IRGLM), Montreal, Quebec, Canada

REFERENCES:
- [Background] Cruccu G, Truini A. A review of Neuropathic Pain: From Guidelines to Clinical Practice. Pain Ther. 2017 Dec;6(Suppl 1):35-42. doi: 10.1007/s40122-017-0087-0. Epub 2017 Nov 24. PMID 29178033
- [Background] Rodrigues L, Moncion K, Eng JJ, Noguchi KS, Wiley E, de Las Heras B, Sweet SN, Fung J, MacKay-Lyons M, Nelson AJ, Medeiros D, Crozier J, Thiel A, Tang A, Roig M. Intensity matters: protocol for a randomized controlled trial exercise intervention for individuals with chronic stroke. Trials. 2022 May 24;23(1):442. doi: 10.1186/s13063-022-06359-w. PMID 35610659
- [Background] Shackleton C, Hodgkiss D, Samejima S, Miller T, Perez MA, Nightingale TE, Sachdeva R, Krassioukov AV. When the whole is greater than the sum of its parts: a scoping review of activity-based therapy paired with spinal cord stimulation following spinal cord injury. J Neurophysiol. 2022 Nov 1;128(5):1292-1306. doi: 10.1152/jn.00367.2022. Epub 2022 Oct 12. PMID 36222423
- [Background] Barthelemy D, Willerslev-Olsen M, Lundell H, Conway BA, Knudsen H, Biering-Sorensen F, Nielsen JB. Impaired transmission in the corticospinal tract and gait disability in spinal cord injured persons. J Neurophysiol. 2010 Aug;104(2):1167-76. doi: 10.1152/jn.00382.2010. Epub 2010 Jun 16. PMID 20554839
- [Background] Barthelemy D, Willerslev-Olsen M, Lundell H, Biering-Sorensen F, Nielsen JB. Assessment of transmission in specific descending pathways in relation to gait and balance following spinal cord injury. Prog Brain Res. 2015;218:79-101. doi: 10.1016/bs.pbr.2014.12.012. Epub 2015 Mar 29. PMID 25890133
- [Background] Megia Garcia A, Serrano-Munoz D, Taylor J, Avendano-Coy J, Gomez-Soriano J. Transcutaneous Spinal Cord Stimulation and Motor Rehabilitation in Spinal Cord Injury: A Systematic Review. Neurorehabil Neural Repair. 2020 Jan;34(1):3-12. doi: 10.1177/1545968319893298. Epub 2019 Dec 20. PMID 31858871
- [Background] Gerasimenko YP, Lu DC, Modaber M, Zdunowski S, Gad P, Sayenko DG, Morikawa E, Haakana P, Ferguson AR, Roy RR, Edgerton VR. Noninvasive Reactivation of Motor Descending Control after Paralysis. J Neurotrauma. 2015 Dec 15;32(24):1968-80. doi: 10.1089/neu.2015.4008. Epub 2015 Aug 20. PMID 26077679
- [Background] Gerasimenko Y, Gorodnichev R, Puhov A, Moshonkina T, Savochin A, Selionov V, Roy RR, Lu DC, Edgerton VR. Initiation and modulation of locomotor circuitry output with multisite transcutaneous electrical stimulation of the spinal cord in noninjured humans. J Neurophysiol. 2015 Feb 1;113(3):834-42. doi: 10.1152/jn.00609.2014. Epub 2014 Nov 5. PMID 25376784
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Background] Inanici F, Samejima S, Gad P, Edgerton VR, Hofstetter CP, Moritz CT. Transcutaneous Electrical Spinal Stimulation Promotes Long-Term Recovery of Upper Extremity Function in Chronic Tetraplegia. IEEE Trans Neural Syst Rehabil Eng. 2018 Jun;26(6):1272-1278. doi: 10.1109/TNSRE.2018.2834339. PMID 29877852
- [Background] Michie S, Johnston M, Abraham C, Lawton R, Parker D, Walker A; "Psychological Theory" Group. Making psychological theory useful for implementing evidence based practice: a consensus approach. Qual Saf Health Care. 2005 Feb;14(1):26-33. doi: 10.1136/qshc.2004.011155. PMID 15692000
- [Background] Brotherton SS, Saunders LL, Krause JS, Morrisette DC. Association between reliance on devices and people for walking and ability to walk community distances among persons with spinal cord injury. J Spinal Cord Med. 2012 May;35(3):156-61. doi: 10.1179/2045772312Y.0000000012. PMID 22507025
- [Background] Laferriere S, Bonizzato M, Cote SL, Dancause N, Lajoie G. Hierarchical Bayesian Optimization of Spatiotemporal Neurostimulations for Targeted Motor Outputs. IEEE Trans Neural Syst Rehabil Eng. 2020 Jun;28(6):1452-1460. doi: 10.1109/TNSRE.2020.2987001. Epub 2020 Apr 13. PMID 32286996
- [Background] Gill ML, Grahn PJ, Calvert JS, Linde MB, Lavrov IA, Strommen JA, Beck LA, Sayenko DG, Van Straaten MG, Drubach DI, Veith DD, Thoreson AR, Lopez C, Gerasimenko YP, Edgerton VR, Lee KH, Zhao KD. Neuromodulation of lumbosacral spinal networks enables independent stepping after complete paraplegia. Nat Med. 2018 Nov;24(11):1677-1682. doi: 10.1038/s41591-018-0175-7. Epub 2018 Sep 24. PMID 30250140
- [Background] Wagner FB, Mignardot JB, Le Goff-Mignardot CG, Demesmaeker R, Komi S, Capogrosso M, Rowald A, Seanez I, Caban M, Pirondini E, Vat M, McCracken LA, Heimgartner R, Fodor I, Watrin A, Seguin P, Paoles E, Van Den Keybus K, Eberle G, Schurch B, Pralong E, Becce F, Prior J, Buse N, Buschman R, Neufeld E, Kuster N, Carda S, von Zitzewitz J, Delattre V, Denison T, Lambert H, Minassian K, Bloch J, Courtine G. Targeted neurotechnology restores walking in humans with spinal cord injury. Nature. 2018 Nov;563(7729):65-71. doi: 10.1038/s41586-018-0649-2. Epub 2018 Oct 31. PMID 30382197
- [Background] Angeli CA, Boakye M, Morton RA, Vogt J, Benton K, Chen Y, Ferreira CK, Harkema SJ. Recovery of Over-Ground Walking after Chronic Motor Complete Spinal Cord Injury. N Engl J Med. 2018 Sep 27;379(13):1244-1250. doi: 10.1056/NEJMoa1803588. Epub 2018 Sep 24. PMID 30247091
- [Background] Hubscher CH, Herrity AN, Williams CS, Montgomery LR, Willhite AM, Angeli CA, Harkema SJ. Improvements in bladder, bowel and sexual outcomes following task-specific locomotor training in human spinal cord injury. PLoS One. 2018 Jan 31;13(1):e0190998. doi: 10.1371/journal.pone.0190998. eCollection 2018. PMID 29385166
- [Background] Evans RW, Shackleton CL, West S, Derman W, Laurie Rauch HG, Baalbergen E, Albertus Y. Robotic Locomotor Training Leads to Cardiovascular Changes in Individuals With Incomplete Spinal Cord Injury Over a 24-Week Rehabilitation Period: A Randomized Controlled Pilot Study. Arch Phys Med Rehabil. 2021 Aug;102(8):1447-1456. doi: 10.1016/j.apmr.2021.03.018. Epub 2021 Apr 9. PMID 33839105
- [Background] Behrman AL, Ardolino EM, Harkema SJ. Activity-Based Therapy: From Basic Science to Clinical Application for Recovery After Spinal Cord Injury. J Neurol Phys Ther. 2017 Jul;41 Suppl 3(Suppl 3 IV STEP Spec Iss):S39-S45. doi: 10.1097/NPT.0000000000000184. PMID 28628595
- [Background] Behrman AL, Bowden MG, Nair PM. Neuroplasticity after spinal cord injury and training: an emerging paradigm shift in rehabilitation and walking recovery. Phys Ther. 2006 Oct;86(10):1406-25. doi: 10.2522/ptj.20050212. PMID 17012645
- [Background] Noonan VK, Fingas M, Farry A, Baxter D, Singh A, Fehlings MG, Dvorak MF. Incidence and prevalence of spinal cord injury in Canada: a national perspective. Neuroepidemiology. 2012;38(4):219-26. doi: 10.1159/000336014. Epub 2012 Apr 27. PMID 22555590